CLINICAL TRIAL: NCT00764686
Title: A Study Investigating an Exercise and Education Programme for Individuals With Ankylosing Spondylitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Ms Anne-Marie Keown, Physiotherapy Manager, Mater Misericordiae University Hospital, Eccles Street, Dublin 7, Ireland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS/2008/83; 1/378/1173
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Spondylitis, Ankylosing
Keywords: Exercise; Education; Hydrotherapy; Physical Therapy Modalities
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Low disease severity group
  Interventions: Other: Exercise and Education
- 2 (Experimental): Higher disease severity group
  Interventions: Other: Exercise and Education

INTERVENTIONS:
Other: Exercise and Education — One hydrotherapy class, one land-exercise class and one education session daily, for five days. Each exercise class and education session is one hour in duration.
  Arms: 2
Other: Exercise and Education — Two hydrotherapy classes, one land-exercise class and one education session daily, for five days. Each exercise class and education are one hour in duration.
  Arms: 1

SUMMARY:
Ankylosing Spondylitis(AS) is a chronic, inflammatory, rheumatic disease (Khan, 2002). AS is associated with increased work disability and use of healthcare resources (Ward et al, 2008). Evidence suggests that group exercise is the most effective form of physiotherapy management for individuals with Ankylosing Spondylitis (Dagfinrud et al, 2008). To date, no research has been published in relation to short, intensive group exercise programmes.

This study aims to investigate the effects of a five day exercise and education programme for individuals with Ankylosing Spondylitis. Effects of the programme on disease activity, function and spinal mobility will be measured using using validated quantitative measures; the overall value of the programme for patients will be explored by means of semi-structured interviews.

DETAILED DESCRIPTION:
Patients with a diagnosis of Ankylosing Spondylitis are referred to the 5-day exercise and education programme by consultant rheumatologists at the Mater Misericordiae University Hospital. All patients referred to the programmes beginning 06/24/2008 and 08/25/2008 will be invited to participate.

Participants scoring 0-6 on the Bath Ankylosing Spondylitis Metrology Index are classified as low disease severity level and are allocated to Group 1; participants with a score of 6.1-10 are classified as higher disease severity and allocated to Group 2. Group 1 has two hydrotherapy classes, a gym-based exercise class and an education session daily. Group 2 has one hydrotherapy class, a gym-based exercise class and an education session daily. Exercise sessions are 1 hour in duration and are given by staff physiotherapists. Education sessions are 1 hour in duration and are given by senior members of the rheumatology multi-disciplinary team at the Mater Misericordiae University Hospital.

Outcome will be assessed upon entry to the study (pre-intervention), at 5 days (post-intervention) and at 4 weeks (follow-up). A semi structured interview will be carried out with each participant immediately post-intervention to explore the overall value of the group programme for participants.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Ankylosing Spondylitis according to the modified New York criteria

Exclusion Criteria:

* Patients for whom hydrotherapy or land-exercise have been contra-indicated
* Cognitive Impairment
* Patients unwilling to give informed, written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Pre-intervention, post-intervention and 4-week follow-up

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Functional Index (BASFI) | Pre-intervention, post intervention and 4-week follow-up
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Pre-intervention, post-intervention and 4-week follow-up.
Semi-structured interview | Post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Keown, BSc MSc, Principal Investigator — Mater Misericordiae University Hospital; Tara Cusack, PhD, Principal Investigator — University College Dublin
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland